CLINICAL TRIAL: NCT00142129
Title: Phase II Study of Velcade in Waldenstrom's Macroglobulinemia
Brief Title: Bortezomib (Velcade) in Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-248
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Waldenstrom's Macroglobulinemia; Lymphoplasmacytic Lymphoma
Keywords: bortezomib; Velcade; Waldenstrom's macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone | interventions — Bortezomib

INTERVENTIONS:
Drug: Bortezomib (Velcade)

SUMMARY:
The purpose of this study is to evaluate how tumors in patients with Waldenstrom's macroglobulinemia respond to treatment with bortezomib (Velcade) and to see what effects (good and bad) it has on the cancer.

DETAILED DESCRIPTION:
* Patients will receive bortezomib intravenously twice weekly for 2 weeks on days 1,4,8 and 11 of each cycle. A 10-day rest period (days 12-21) will follow the 2 weeks of treatment. The treatment cycle is repeated up to eight times depending upon the disease response and if the patient is tolerating the drugs.
* The following procedures will be conducted as part of the treatment monitoring: DAY 1 VISIT (of each treatment cycle): evaluation of disease-related symptoms, vital signs and weight and blood tests. DAY 4 VISIT (of each treatment cycle): vital signs and blood work. DAY 8 VISIT (of each treatment cycle): vital signs and blood work. DAY 11 VISIT(of each treatment cycle): vital signs, blood work, and possible CT Scan.
* Treatment will be discontinued if any of the following occur: Disease gets worse, severe side-effects or the patient requires other anti-cancer therapy.
* At the end of the treatment (30 days after the last dose of study drug) the patient will have a physical exam, vital signs, evaluation of disease-related symptoms, blood work and CT scan for tumor measurements.
* Long term follow-up consists of every 3 month clinical visits until disease progression or up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Clinicopathological diagnosis of Waldenstrom's macroglobulinemia who have failed one first line therapy
* Measurable disease, defined as presence of immunoglobulin M (Ig M) paraprotein with a minimum IgM level of >2 times ULN
* Karnofsky performance status of >60
* Life expectancy of > 3 months
* Baseline platelet count >50,000,000,000/L and ANC of 750,000,000/L
* AST and ALT < 3 x ULN
* Total bilirubin < 2 x ULN
* Calculated or measured creatinine clearance > 30mL/minute
* Serum sodium > 130 mmol/L

Exclusion Criteria:

* Greater than or equal to Grade 2 peripheral neuropathy
* Hypersensitivity to bortezomib, boron or mannitol
* Prior therapy with Velcade
* Pregnant or lactating women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27
Dates: Start 2003-12; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To determine response rate along with attainment of stable disease following treatment with bortezomib in patients with Waldenstrom's macroglobulinemia.

SECONDARY OUTCOMES:
To assess the safety and tolerability of bortezomib in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Treon, MD, MA, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts